CLINICAL TRIAL: NCT03987243
Title: Mobile and Remote Monitoring of Seating Pressure for Wheelchair Users With SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Minnesota (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Melissa M. Morrow, Ph.D., Associate Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-007531; 1R21AG050640-01A1 (NIH)
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injury; Seating Pressure Mapping; Pressure Injury Prevention; Seating Interface Pressure; Wheelchair User
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This is a longitudinal, within-subject, repeated (A-B-A-B) measures design. Two interventions will be provided: structured education regarding pressure ulcer prevention through weight shifts at start of study and use of a mobile seat interface pressure map (IPM).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Two interventions will be provided. The first intervention is a structured education regarding pressure ulcer prevention through weight shifts at start of study. The second intervention is the use of a mobile seat interface pressure map (IPM), which will occur during two intervention phases.
  Interventions: Behavioral: Structured Pressure Ulcer Prevention Education; Other: Mobile Seat Interface Pressure Mapping System (IPM)

INTERVENTIONS:
Behavioral: Structured Pressure Ulcer Prevention Education — Structured education for performance weight shift maneuvers and pressure ulcer prevention will occur during the initial visit for each subject. The education method used aligns with principles of the social cognitive theory to facilitate learning. The purpose in providing the education is to ensure all of the participants receive uniform instruction in how to perform weight shifts and to facilitate understanding of the importance of completing them as a protective measure against pressure ulcer development. Because each participant will come into the study at varying levels of understanding about pressure ulcer risk and knowledge of how to complete weight shift maneuvers, the education component is critical to ensure all participants are provided with the same information in the same way.
Other: Mobile Seat Interface Pressure Mapping System (IPM) — This mobile IPM system was designed to provide visual information about seat interface pressure distribution to compensate for lack of sensation on the sitting surface. This variable will be toggled on and off between the intervention and control phases of the study. The participants will have access to the visual feedback while learning how to complete weight shift maneuvers at the initial visit and then again at home during the intervention phases (weeks 2 and 4). During the control phases (weeks 1 and 3), they will not have access to the visual feedback from the pressure map

SUMMARY:
This study will examine two interventions to increase weight shifts, overall trunk movement, and self-efficacy related to pressure ulcer prevention in wheelchair users with a spinal cord injury (SCI).

DETAILED DESCRIPTION:
Participants will use a mobile seat interface pressure mapping system that gives them live, real-time, visual feedback on the distribution of pressure between them and their seat cushion. This type of feedback works as a compensatory strategy for lack of sensation and allows the individual to visually observe pressure distribution they are not able to feel. Additionally, the participants will be provided with structured pressure ulcer prevention education, grounded in the principles of social cognitive theory, regarding pressure ulcer risk and use of weight shifts.

The pressure mapping system, which will be used during training, provides virtual modeling of the desired outcome (reduced pressure) and is an important part of the education module.

The findings of this study will inform clinicians and investigators of whether use of mobile seat interface pressure mapping as a compensatory-based intervention has a positive impact on trunk movement and self-efficacy for completing weight shifts in wheelchair users who lack sensation. Another contribution of this work is an exploration of the relationship between self-efficacy and movement in wheelchair users.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a spinal cord injury (C4 and below, traumatic or non-traumatic, with onset greater than 12 months at enrollment)
* Individuals who use a wheelchair as their primary form of mobility
* Individuals who are willing to participate and able to make 2 visits to the Mayo Clinic in Rochester, MN

Exclusion Criteria:

* Documented active pressure ulcer of any stage at initiation of study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Trunk Movement | For each phase and session combination (A1, B1, A2, B2), the daily values will be averaged over the 7 day collection period for one representative daily percentage of trunk active movement.
  The primary outcome variable, trunk movement, will be defined by the percentage of the day with active trunk movement.

SECONDARY OUTCOMES:
Total Vector Magnitude of Movement | For each phase and session combination (A1, B1, A2, B2), the daily values will be averaged over the 7 day collection period for one representative daily percentage of trunk active movement.
  The vector magnitude for each second of data during wear-times will be classified as a period of activity or inactivity.
Forward and Lateral Tilt | For each phase and session combination (A1, B1, A2, B2), the daily values will be averaged over the 7 day collection period for one representative daily percentage of trunk active movement.
  Forward and lateral tilt will be assessed with the raw triaxial accelerometer data by determining the angles between gravity and the off-axes

CONTACTS AND LOCATIONS:
Overall Officials: Melissa MB Morrow, PhD, Principal Investigator — Mayo Clinic; Tamara L Vos-Draper, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krause JS. Skin sores after spinal cord injury: relationship to life adjustment. Spinal Cord. 1998 Jan;36(1):51-6. doi: 10.1038/sj.sc.3100528. PMID 9471139
- [Background] Raghavan P, Raza WA, Ahmed YS, Chamberlain MA. Prevalence of pressure sores in a community sample of spinal injury patients. Clin Rehabil. 2003 Dec;17(8):879-84. doi: 10.1191/0269215503cr692oa. PMID 14682560
- [Background] Fuhrer MJ, Garber SL, Rintala DH, Clearman R, Hart KA. Pressure ulcers in community-resident persons with spinal cord injury: prevalence and risk factors. Arch Phys Med Rehabil. 1993 Nov;74(11):1172-7. PMID 8239957
- [Background] Akins JS, Karg PE, Brienza DM. Interface shear and pressure characteristics of wheelchair seat cushions. J Rehabil Res Dev. 2011;48(3):225-34. doi: 10.1682/jrrd.2009.09.0145. PMID 21480097
- [Background] Bates-Jensen BM, Guihan M, Garber SL, Chin AS, Burns SP. Characteristics of recurrent pressure ulcers in veterans with spinal cord injury. J Spinal Cord Med. 2009;32(1):34-42. doi: 10.1080/10790268.2009.11760750. PMID 19264047
- [Background] Mawson AR, Biundo JJ Jr, Neville P, Linares HA, Winchester Y, Lopez A. Risk factors for early occurring pressure ulcers following spinal cord injury. Am J Phys Med Rehabil. 1988 Jun;67(3):123-7. doi: 10.1097/00002060-198806000-00007. PMID 3377890
- [Background] Niazi ZB, Salzberg CA, Byrne DW, Viehbeck M. Recurrence of initial pressure ulcer in persons with spinal cord injuries. Adv Wound Care. 1997 May-Jun;10(3):38-42. PMID 9306777
- [Background] Staas WE Jr, Cioschi HM. Pressure sores--a multifaceted approach to prevention and treatment. West J Med. 1991 May;154(5):539-44. PMID 1830985
- [Background] Thomas DR. Prevention and treatment of pressure ulcers: what works? what doesn't? Cleve Clin J Med. 2001 Aug;68(8):704-7, 710-14, 717-22. doi: 10.3949/ccjm.68.8.704. PMID 11510528
- [Background] Thietje R, Giese R, Pouw M, Kaphengst C, Hosman A, Kienast B, van de Meent H, Hirschfeld S. How does knowledge about spinal cord injury-related complications develop in subjects with spinal cord injury? A descriptive analysis in 214 patients. Spinal Cord. 2011 Jan;49(1):43-8. doi: 10.1038/sc.2010.96. Epub 2010 Sep 7. PMID 20820180
- [Background] Verschueren JH, Post MW, de Groot S, van der Woude LH, van Asbeck FW, Rol M. Occurrence and predictors of pressure ulcers during primary in-patient spinal cord injury rehabilitation. Spinal Cord. 2011 Jan;49(1):106-12. doi: 10.1038/sc.2010.66. Epub 2010 Jun 8. PMID 20531357
- [Background] Consortium for Spinal Cord Medicine Clinical Practice Guidelines. Pressure ulcer prevention and treatment following spinal cord injury: a clinical practice guideline for health-care professionals. J Spinal Cord Med. 2001 Spring;24 Suppl 1:S40-101. doi: 10.1080/10790268.2001.11753592. No abstract available. PMID 11958176
- [Background] Clark FA, Jackson JM, Scott MD, Carlson ME, Atkins MS, Uhles-Tanaka D, Rubayi S. Data-based models of how pressure ulcers develop in daily-living contexts of adults with spinal cord injury. Arch Phys Med Rehabil. 2006 Nov;87(11):1516-25. doi: 10.1016/j.apmr.2006.08.329. PMID 17084129
- [Background] Dunn CA, Carlson M, Jackson JM, Clark FA. Response factors surrounding progression of pressure ulcers in community-residing adults with spinal cord injury. Am J Occup Ther. 2009 May-Jun;63(3):301-9. doi: 10.5014/ajot.63.3.301. PMID 19522138
- [Background] Stinson MD, Porter-Armstrong AP, Eakin PA. Pressure mapping systems: reliability of pressure map interpretation. Clin Rehabil. 2003 Aug;17(5):504-11. doi: 10.1191/0269215503cr643oa. PMID 12952156
- [Background] Crawford SA, Strain B, Gregg B, Walsh DM, Porter-Armstrong AP. An investigation of the impact of the Force Sensing Array pressure mapping system on the clinical judgement of occupational therapists. Clin Rehabil. 2005 Mar;19(2):224-31. doi: 10.1191/0269215505cr826oa. PMID 15759539
- [Background] Norman D. Measuring interface pressure: validity and reliability problems. J Wound Care. 2004 Feb;13(2):78-80. doi: 10.12968/jowc.2004.13.2.26576. PMID 14999994
- [Background] Sprigle S, Sonenblum S. Assessing evidence supporting redistribution of pressure for pressure ulcer prevention: a review. J Rehabil Res Dev. 2011;48(3):203-13. doi: 10.1682/jrrd.2010.05.0102. PMID 21480095
- [Background] Brienza DM, Karg PE, Geyer MJ, Kelsey S, Trefler E. The relationship between pressure ulcer incidence and buttock-seat cushion interface pressure in at-risk elderly wheelchair users. Arch Phys Med Rehabil. 2001 Apr;82(4):529-33. doi: 10.1053/apmr.2001.21854. PMID 11295017
- [Background] Stinson M, Porter A, Eakin P. Measuring interface pressure: a laboratory-based investigation into the effects of repositioning and sitting. Am J Occup Ther. 2002 Mar-Apr;56(2):185-90. doi: 10.5014/ajot.56.2.185. PMID 11905303
- [Background] Barnett RI, Shelton FE 4th. Measurement of support surface efficacy: pressure. Adv Wound Care. 1997 Nov-Dec;10(7):21-9. Erratum In: Adv Wound Care 1998 Mar-Apr;11(2):94. PMID 9450403
- [Background] Bogie K, Wang X, Fei B, Sun J. New technique for real-time interface pressure analysis: getting more out of large image data sets. J Rehabil Res Dev. 2008;45(4):523-35, 10 p following 535. doi: 10.1682/jrrd.2007.03.0046. PMID 18712638
- [Background] Crawford SA, Stinson MD, Walsh DM, Porter-Armstrong AP. Impact of sitting time on seat-interface pressure and on pressure mapping with multiple sclerosis patients. Arch Phys Med Rehabil. 2005 Jun;86(6):1221-5. doi: 10.1016/j.apmr.2004.08.010. PMID 15954063
- [Background] Eitzen I. Pressure mapping in seating: a frequency analysis approach. Arch Phys Med Rehabil. 2004 Jul;85(7):1136-40. doi: 10.1016/j.apmr.2003.09.007. PMID 15241764
- [Background] Reenalda J, Jannink M, Nederhand M, IJzerman M. Clinical use of interface pressure to predict pressure ulcer development: a systematic review. Assist Technol. 2009 Summer;21(2):76-85. doi: 10.1080/10400430903050437. PMID 19715252
- [Background] Jackson J, Carlson M, Rubayi S, Scott MD, Atkins MS, Blanche EI, Saunders-Newton C, Mielke S, Wolfe MK, Clark FA. Qualitative study of principles pertaining to lifestyle and pressure ulcer risk in adults with spinal cord injury. Disabil Rehabil. 2010;32(7):567-78. doi: 10.3109/09638280903183829. PMID 20136475
- [Background] Pipkin L, Sprigle S. Effect of model design, cushion construction, and interface pressure mats on interface pressure and immersion. J Rehabil Res Dev. 2008;45(6):875-82. doi: 10.1682/jrrd.2007.06.0089. PMID 19009473
- [Background] Saunders LL, Krause JS, Acuna J. Association of race, socioeconomic status, and health care access with pressure ulcers after spinal cord injury. Arch Phys Med Rehabil. 2012 Jun;93(6):972-7. doi: 10.1016/j.apmr.2012.02.004. Epub 2012 Apr 10. PMID 22494948
- [Background] Stinson M, Schofield R, Gillan C, Morton J, Gardner E, Sprigle S, Porter-Armstrong A. Spinal cord injury and pressure ulcer prevention: using functional activity in pressure relief. Nurs Res Pract. 2013;2013:860396. doi: 10.1155/2013/860396. Epub 2013 Apr 9. PMID 23691301
- [Background] Maurer CL, Sprigle S. Effect of seat inclination on seated pressures of individuals with spinal cord injury. Phys Ther. 2004 Mar;84(3):255-61. PMID 14984297
- [Background] Sprigle S, Dunlop W, Press L. Reliability of bench tests of interface pressure. Assist Technol. 2003 Summer;15(1):49-57. doi: 10.1080/10400435.2003.10131889. PMID 14760981
- [Background] Fortune E, Lugade V, Morrow M, Kaufman K. Validity of using tri-axial accelerometers to measure human movement - Part II: Step counts at a wide range of gait velocities. Med Eng Phys. 2014 Jun;36(6):659-69. doi: 10.1016/j.medengphy.2014.02.006. Epub 2014 Mar 20. PMID 24656871
- [Background] Lugade V, Fortune E, Morrow M, Kaufman K. Validity of using tri-axial accelerometers to measure human movement - Part I: Posture and movement detection. Med Eng Phys. 2014 Feb;36(2):169-76. doi: 10.1016/j.medengphy.2013.06.005. Epub 2013 Jul 27. PMID 23899533
- [Derived] Vos-Draper TL, Morrow MMB, Ferguson JE, Mathiowetz VG. Effects of Real-Time Pressure Map Feedback on Confidence in Pressure Management in Wheelchair Users With Spinal Cord Injury: Pilot Intervention Study. JMIR Rehabil Assist Technol. 2023 Oct 12;10:e49813. doi: 10.2196/49813. PMID 37824188
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT03987243/Prot_SAP_000.pdf